CLINICAL TRIAL: NCT05494879
Title: Evaluation of the Effect of Microkinesitherapy Treatment on Psychosomatic Functions in Community-dwelling Older Adults: A Pilot Study
Brief Title: Effectiveness of Microkinesitherapy in Seniors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Opole University of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Micro_Poznan
Record Dates: First submitted 2022-07-29; First posted 2022-08-10 (Actual); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Microkinesitherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- microkinesitherapy treatment (Experimental): The study group received a single therapy session of microkinesitherapy. The entire procedure lasted about 10 minutes. Microkinesitherapy is based on locating information in the patient's body about previous traumas/traumas that have been experienced physically and emotionally, which the body could not eliminate. This information is interpreted on the body by sensitive tensions and called "body scars" and does not necessarily remain in the brain.
  Interventions: Behavioral: microkinesitherapy treatment

INTERVENTIONS:
Behavioral: microkinesitherapy treatment — The therapeutic session of microkinesitherapy included a seeking of "body scares" both taking into account somatic dysfunctions as well as psychosomatic disorders. According to the creators of the method, Grosjean and Benini "Everything that happens with us in a toxic level, either physically or emotionally, are stored by the brain which keeps memories and generates links that may harm the function of the cells generating a vast array of symptoms and dysfunctions".

SUMMARY:
Many specialists stress that the aging process is individual, its course, severity and occurrence of disease are not the same for all seniors. The studies indicate that SA should be conceptualized as a process, using developmental trajectories of functioning as component parts, and can take several forms. The nature of "successful" trajectories varied from a limited decline over time (e.g., cognitive and physical functioning), stability over time (e.g., self-perceived health) to recovery (from social loneliness) and growth (in life satisfaction and emotional support provided). Therefore, the aim of this study was to investigate the effectiveness of microkinesitherapy treatment in community-dwelling older adults.

DETAILED DESCRIPTION:
new therapeutic methods are being proposed that can be used in the community to steer the aging process toward "healthy aging." An example of a holistic approach to the patient can be found in microkinesitherapy. The focus of microkinesitherapy is to find and restore areas of the body that have lost their vitality and mobility, using gentle touches on various body tissues using specific body maps. The aim of this study was to investigate the effectiveness of microkinesitherapy treatment in community-dwelling older adults. It was decided to evaluate the impact of a single therapy session on a range of psycho-somatic indicators. The hypotheses were as follows: (H1) The microkinesitherapy intervention will improve the physical function assessed using the Senior Fitness Test, (H2) A single microkinesitherapy treatment will not affect gait performance, (H3) A single microkinesitherapy treatment will improve the quality of life of the participants.

ELIGIBILITY:
Inclusion Criteria:

* informed consent to participate in the study

Exclusion Criteria:

* pneumonia, tuberculosis and other respiratory inflammatory disease in all stages and forms
* less than 6 months after a heart attack, state after thoracic and cardiac surgery
* uncontrolled hypertension
* insulin-dependent diabetes
* lung cancer
* cognitive impairment or Mini-Mental State Examination < 24.

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-08-17 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2023-07-18 (Estimated)

PRIMARY OUTCOMES:
Change of the Senior Fitness Test | baseline, 1-month follow-up
  The Senior Fitness Test (also known as the Fullerton test) was used to assess physical fitness. Five motor tasks were evaluated, including strength, endurance, flexibility, agility, balance, and motor coordination. The sixth component of the test: the 6-minute walk test could not be performed due to the patients' low functional status.
Change of the gait parameters | baseline, 1-month follow-up
  Gait cycle analysis was performed with the subject barefoot over a distance of 5 m long and 2 m wide, making 2 passes (10 m) at normal gait speed. For gait analysis, a wireless inertial sensor system BTS G-WALK (BTS Bioengineering S.p.A., Milan, Italy) was used, placed by means of a semi-elastic belt at the level of the fifth lumbar vertebra (L5) and the first two sacral vertebrae (S1-S2).
Change of the quality of life | baseline, 1-month follow-up
  The WHO's questions stem from multiple statements about quality of life, health and well-being from people with and without disease, and health professionals. The questionnaire was validated and identifies four major domains: Physical health, Psychological, Social relationships, Environment. Each individual item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale. The scores are then transformed to a 0-100 or 4-20 scales. Lower score indicates poorer quality of life
Change of the mental health | baseline, 1-month follow-up
  The GHQ-12 General Health Questionnaire enables the identification of people whose mental state has broken down temporarily or over the long term as a result of difficulties experienced, problems or as a result of mental illness, and those who are at significant risk of mental health disorders. A version of the GHQ-28 provides an overall score that is an indicator of the patient's mental health, divided into 4 scales: somatic symptoms; anxiety, insomnia; dysfunction and symptoms of depression. The scoring type used in this study was Likert scoring methods (0-1-2-3). Higher score indicates greater disorder

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physical Education and Physiotherapy, Opole University of Technology, Opole, Poland

IPD SHARING:
Plan to Share IPD: Yes
The data presented in this study are available upon request from the corresponding author.
Supporting Information: Study Protocol
Time Frame: 6-months